CLINICAL TRIAL: NCT07357051
Title: A Multicenter, Randomized, Double-blind, Double-dummy, Active-controlled Phase III Clinical Study Evaluating the Safety, Pharmacokinetics, and Efficacy of JKN2301 Dry Suspension in Pediatric Patients Aged 2 to Under 12 Years With Influenza
Brief Title: Phase III Clinical Study Evaluating the Safety, Pharmacokinetics, and Efficacy of JKN2301 Dry Suspension in Pediatric Patients Aged 2 to Under 12 Years With Influenza
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Joincare Pharmaceutical Group Industry Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JKN2301-III-01
Record Dates: First submitted 2026-01-08; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Viral Infection
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JKN2301 + Oseltamivir Placebo (Experimental)
  Interventions: Drug: JKN2301 Dry Suspension; Drug: Oseltamivir Placebo
- Oseltamivir + JKN2301 Placebo (Active Comparator)
  Interventions: Drug: Oseltamivir; Drug: JKN2301 Placebo

INTERVENTIONS:
Drug: JKN2301 Dry Suspension — Single oral dose, administered according to a weight-tiered dosing scheme.
  Arms: JKN2301 + Oseltamivir Placebo
Drug: Oseltamivir Placebo — Oral suspension, administered twice daily for 5 days, matched to the weight-based dosing of active oseltamivir.
  Arms: JKN2301 + Oseltamivir Placebo
Drug: Oseltamivir — Oral suspension, administered twice daily for 5 days according to the approved weight-based dosing regimen.
  Arms: Oseltamivir + JKN2301 Placebo
Drug: JKN2301 Placebo — Single oral dose, matched to the weight-tiered dosing scheme of active JKN2301.
  Arms: Oseltamivir + JKN2301 Placebo

SUMMARY:
The goal of this phase III study is to learn if JKN2301 Dry Suspension works to treat uncomplicated influenza in Pediatric Participants aged 2 to 11 years.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients within the specified age range.
* Clinical presentation consistent with influenza, confirmed by a positive local rapid test or central laboratory PCR test.
* Presentation for treatment within the early symptomatic phase of influenza illness.
* Presence of fever and at least one respiratory symptom.
* Ability to swallow oral suspension.
* Parent/guardian and patient (as age-appropriate) able to provide informed consent/assent.

Exclusion Criteria:

* Clinical signs suggestive of severe or complicated influenza infection
* requiring inpatient management.
* Presence of a concurrent bacterial infection requiring systemic therapy.
* Significant immunocompromised, or severe/uncontrolled comorbid conditions.
* History of hypersensitivity to any component of the investigational products.
* Use of prohibited medications (including other anti-influenza antivirals) within a specified period prior to enrollment.
* Recent participation in another interventional clinical trial.
* Any condition that, in the opinion of the investigator, would jeopardize patient safety or compliance with the study protocol.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and relationship to treatment of adverse events (AEs) and serious adverse events (SAEs) | Baseline through Day 15
Clinically significant changes in laboratory parameters, vital signs, physical examination, and ECG | Baseline through Day 15

SECONDARY OUTCOMES:
Plasma concentration-time profiles of JKN2301 and its relevant metabolites | At multiple timepoints up to Day 6
Time to alleviation of all influenza symptoms | From treatment initiation up to Day 15
Duration of fever | From treatment initiation up to Day 15
Time to cessation of viral shedding assessed by viral culture | From treatment initiation up to Day 9
Change from baseline in viral titer | Baseline to Day 9
Incidence of influenza-related complications | Up to Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China